CLINICAL TRIAL: NCT00957359
Title: Effects of Psilocybin on Anxiety and Psychosocial Distress in Cancer Patients
Brief Title: Psilocybin Cancer Anxiety Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-954
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Cancer
Keywords: Cancer; Anxiety; Depression; Hallucinogens
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression | interventions — Psilocybin; Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin (Experimental): Drug intervention
  Interventions: Drug: Psilocybin; Drug: Niacin
- Niacin (Active Comparator): Active control
  Interventions: Drug: Psilocybin; Drug: Niacin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin is a serotonergic hallucinogen that will be administered once at a dose of 0.3mg/kg
  Other Names: 4-phosphoryloxy-N,N-dimethyltryptamine
Drug: Niacin — Psilocybin and niacin will be administered in identically appearing opaque, size 0 gelatin capsules with approximately 180ml of water. The niacin dose will be 250mg

SUMMARY:
The primary objective of this double-blind, placebo-controlled pilot study is to assess the efficacy of psilocybin administration (4-phosphoryloxy-N,N-dimethyltryptamine), a serotonergic psychoactive agent, on psychosocial distress, with the specific primary outcome variable being anxiety associated with cancer. Secondary outcome measures will look at the effect of psilocybin on symptoms of pain perception, depression, existential/psychospiritual distress, attitudes towards disease progression and death, quality of life, and spiritual/mystical states of consciousness. In addition, a secondary objective of the study is to determine the feasibility of administering psilocybin to this patient population, with regards to the following issues: safety, patient recruitment, consent for treatment, and retention. The duration of the proposed investigation will be long enough to administer the drug one time to each of thirty-two patients and to conduct follow-up assessments. This study is separate but similar to a recently completed study at the Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, run by a psychiatrist, Dr. Charles Grob. Although the outcomes measures would be similar to those used as in the Grob study, the proposed dose of psilocybin is higher at 0.3mg/kg and the total subjects for the study would be 32 instead of 12. The study utilizes a cross-over design at 7 weeks and includes prospective follow-up of 6 months duration. This study has been approved by the Bellevue Psychiatry Research Committee, the NYU Oncology PRMC Committee, the Food and Drug Administration (FDA) through the issuance of an IND (77,138), the New York University School of Medicine Institutional Review Board (NYU IRB), the Health and Hospitals Corporation (HHC)-New York University (NYU) Clinical Translational Science Institute (CTSI), the NYU Bluestone Center for Clinical Research, and the Drug Enforcement Agency (DEA) through the issuance of a schedule I license.

It is hypothesized that a one time experience with psilocybin will occasion dramatic shifts in consciousness and awareness that will lead to short-term (ie hours to days) and long-term (up to 6 months in this study, following the administration of the second dosing, either psilocybin or placebo) improvement in anxiety, depression, and pain associated with advanced cancer. The exact mechanism of action is unclear but based on studies done in the 60's using serotonergic hallucinogens in patients with advanced cancer, improvements in anxiety levels, mood and pain were reported. However, a treatment model developed by the famous British psychiatrist Humphrey Osmond, offers one possibility. In this model, serotonergic hallucinogens' therapeutic mechanism lies in their ability to allow the individual to access novel dimensions of consciousness and their efficacy or lack thereof relies on whether a transcendent and mystical state of awareness is attained. Another possible mechanism relates to what Dobkin de Rios and Grob have described as 'managed altered states of consciousness,' where the power of suggestibility, occurring in a safe setting, allows one to transcend a particular state of consciousness (i.e. anxiety and depression associated with advanced illness) as a means to facilitate emotional discharge and to manage irreconcilable conflict.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-76
* Current or historical diagnosis of cancer
* Projected life expectancy of at least one year
* DSM-IV diagnoses: Acute Stress Disorder, Generalized Anxiety Disorder, Anxiety Disorder due to cancer, Adjustment Disorder with anxious features
* Any stage of cancer diagnosis

Exclusion Criteria:

* Epilepsy
* Renal disease
* Diabetes
* Abnormal liver function
* Severe cardiovascular disease
* Malignant Hypertension
* Baseline blood pressure must be less than or equal to 140/90
* Personal history or immediate family members with schizophrenia, bipolar affective disorder, delusional disorder, schizoaffective disorder or other psychotic spectrum illness
* Current substance use disorder
* Medication contraindications: anti-seizures medications, insulin, oral hypoglycemics, clonidine, aldomet, cardiovascular medications, anti-psychotics (first and second generation), anti-depressants and mood stabilizers

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ross, MD, Principal Investigator — NYU Langone Health; Anthony Bossis, PhD, Study Chair — Co-Principal Investigator NYU Langone School of Medicine; Jeffrey Guss, MD, Study Director — Co-Principal Investigator NYU Langone School of Medicine
Locations (1):
- NYU College of Dentistry Bluestone Center for Clinical Research, New York, New York, United States

REFERENCES:
- [Derived] Agin-Liebes GI, Malone T, Yalch MM, Mennenga SE, Ponte KL, Guss J, Bossis AP, Grigsby J, Fischer S, Ross S. Long-term follow-up of psilocybin-assisted psychotherapy for psychiatric and existential distress in patients with life-threatening cancer. J Psychopharmacol. 2020 Feb;34(2):155-166. doi: 10.1177/0269881119897615. Epub 2020 Jan 9. PMID 31916890
- [Derived] Ross S, Bossis A, Guss J, Agin-Liebes G, Malone T, Cohen B, Mennenga SE, Belser A, Kalliontzi K, Babb J, Su Z, Corby P, Schmidt BL. Rapid and sustained symptom reduction following psilocybin treatment for anxiety and depression in patients with life-threatening cancer: a randomized controlled trial. J Psychopharmacol. 2016 Dec;30(12):1165-1180. doi: 10.1177/0269881116675512. PMID 27909164
- See also: Related Info — http://www.nyucanceranxiety.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Psilocybin First, Then Niacin; Niacin First, Then Psilocybin: Psilocybin and niacin will be administered in identically appearing opaque, size 0 gelatin capsules with approximately 180ml of water. The niacin dose will be 250mg.
Period: Overall Study
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Psilocybin First, Then Niacin: Psilocybin: Psilocybin is a serotonergic hallucinogen that will be administered once at a dose of 0.3mg/kg
- Niacin First, Then Psilocybin: Niacin: Psilocybin and niacin will be administered in identically appearing opaque, size 0 gelatin capsules with approximately 180ml of water. The niacin dose will be 250mg
- Total: Total of all reporting groups
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age | 52 (15.03) | 60.27 (9.45) | 56.28 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 7 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: HADS Anxiety
Description: Hospital Anxiety and Depression Scale (HADS) used for measuring anxiety; Scored on a scale of 0-21 (higher score more anxiety)
Time Frame: 2-4 weeks prior to drug administration
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Psilocybin First, Then Niacin: Drug intervention
  Psilocybin: Psilocybin is a serotonergic hallucinogen that will be administered once at a dose of 0.3mg/kg
  Niacin: Psilocybin and niacin will be administered in identically appearing opaque, size 0 gelatin capsules with approximately 180ml of water. The niacin dose will be 250mg
- Niacin First, Then Psilocybin: Active control
  Psilocybin: Psilocybin is a serotonergic hallucinogen that will be administered once at a dose of 0.3mg/kg
  Niacin: Psilocybin and niacin will be administered in identically appearing opaque, size 0 gelatin capsules with approximately 180ml of water. The niacin dose will be 250mg
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 15.14 (1.88) | 16.93 (1.81)

2. Primary Outcome: HADS Anxiety
Description: as for outcome 1
Time Frame: 1 day prior to drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 9.0 (.83) | 9.0 (0.8)

3. Primary Outcome: HADS Anxiety
Description: as for outcome 1
Time Frame: 1 day post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 3.43 (.83) | 6.0 (.80)

4. Primary Outcome: HADS Anxiety
Description: as for outcome 1
Time Frame: 6 weeks post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 4.64 (.83) | 8.44 (.82)

5. Primary Outcome: HADS Anxiety
Description: as for outcome 1
Time Frame: 1 day prior to drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 4.57 (0.88) | 7.98 (0.83)

6. Primary Outcome: HADS Anxiety
Description: as for outcome 1
Time Frame: 6 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 3.60 (.90) | 5.54 (.89)

7. Primary Outcome: HADS Anxiety
Description: as for outcome 1
Time Frame: 26 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 2.69 (.92) | 4.70 (.89)

8. Primary Outcome: State-Trait Anxiety Inventory (STAI) State
Description: STAI scores 20-80 (higher score more anxiety). Commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
Time Frame: 2-4 weeks prior to drug administration/ Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 43.79 (2.83) | 48.53 (2.12)

9. Primary Outcome: STAI State
Description: as for outcome 8
Time Frame: 1 day prior to drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 39.07 (2.83) | 45.6 (2.73)

10. Primary Outcome: STAI State
Description: as for outcome 8
Time Frame: 1 day post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 27.5 (2.83) | 40.33 (2.73)

11. Primary Outcome: HADS Depression
Description: 0-21 (higher score more depression)
Time Frame: 2-4 weeks prior to drug administration/ Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 5.29 (0.92) | 7 (0.89)

12. Primary Outcome: STAI State
Description: as for outcome 8
Time Frame: 6 weeks post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 33.5 (2.83) | 47.05 (2.80)

13. Primary Outcome: STAI State
Description: as for outcome 8
Time Frame: 1 day prior to drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 32.72 (2.99) | 45.31 (2.82)

14. Primary Outcome: STAI State
Description: as for outcome 8
Time Frame: 1 day post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 25.73 (3.04) | 38.11 (2.83)

15. Primary Outcome: STAI State
Description: as for outcome 8
Time Frame: 6 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 30.67 (3.05) | 37.77 (3.07)

16. Primary Outcome: STAI State
Description: as for outcome 8
Time Frame: 26 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 28.04 (3.15) | 38.28 (3.04)

17. Primary Outcome: STAI Trait
Description: as for outcome 8
Time Frame: 2-4 weeks prior to drug administration/ Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 43.79 (2.83) | 48.53 (2.12)

18. Primary Outcome: STAI Trait
Description: as for outcome 8
Time Frame: 1 day prior to drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 39.07 (2.83) | 45.87 (2.12)

19. Primary Outcome: STAI Trait
Description: as for outcome 8
Time Frame: 1 day post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 27.5 (2.83) | 44 (2.12)

20. Primary Outcome: STAI Trait
Description: as for outcome 8
Time Frame: 6 weeks post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 33.5 (2.83) | 46.19 (2.17)

21. Primary Outcome: STAI Trait
Description: as for outcome 8
Time Frame: 1 day prior to drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 32.72 (2.99) | 45.31 (2.82)

22. Primary Outcome: STAI Trait
Description: as for outcome 8
Time Frame: 1 day post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 25.73 (3.04) | 38.11 (2.83)

23. Primary Outcome: STAI Trait
Description: as for outcome 8
Time Frame: 6 weeks prior to drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 30.67 (3.05) | 37.77 (3.07)

24. Primary Outcome: STAI Trait
Description: as for outcome 8
Time Frame: 6 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 28.04 (3.15) | 38.28 (3.04)

25. Primary Outcome: HADS Depression
Description: 0-21 (higher score more depression)
Time Frame: 1 day prior to drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 10.43 (1.88) | 16.47 (1.81)

26. Primary Outcome: HADS Depression
Description: Hospital Anxiety and Depression Scale (HADS) used for measuring depression; Scored on a scale of 0-21 (higher score more depression)
Time Frame: 1 day post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 4.21 (1.88) | 12.07 (1.81)

27. Primary Outcome: HADS Depression
Description: as for outcome 26
Time Frame: 6 weeks post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 6.5 (1.88) | 14.24 (1.84)

28. Primary Outcome: HADS Anxiety
Description: 0-21 (higher score more anxiety)
Time Frame: 1 day post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 6.84 (0.69) | 13.02 (1.85)

29. Primary Outcome: HADS Depression
Description: as for outcome 26
Time Frame: 1 day post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 5.25 (1.97) | 10.05 (1.86)

30. Primary Outcome: HADS Depression
Description: as for outcome 26
Time Frame: 6 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 6.31 (1.99) | 9.65 (1.95)

31. Primary Outcome: HADS Depression
Description: as for outcome 26
Time Frame: 26 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 6.48 (2.04) | 9.06 (1.97)

32. Secondary Outcome: Death Anxiety Scale
Description: 0-15 (higher score more death anxiety)
Time Frame: 26 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 6.71 (0.72) | 6.83 (0.69)

33. Secondary Outcome: Death Anxiety Scale
Description: 0-15 (higher score more death anxiety)
Time Frame: 2 weeks post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 6.57 (0.67) | 7.85 (0.66)

34. Secondary Outcome: Death Transcendence Scale
Description: 0-60 (higher score more death transcendence)
Time Frame: 2-4 weeks prior to drug administration/ Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 13.64 (5.96) | 11.27 (5.76)

35. Secondary Outcome: Hopelessness
Description: 0-16 (higher score more hopeless)
Time Frame: Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 5.71 (0.76) | 6.73 (0.74)

36. Secondary Outcome: Death Anxiety Scale
Description: 0-15 (higher score more death anxiety)
Time Frame: 2-4 weeks prior to drug administration/ Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 9.14 (0.67) | 8.13 (0.64)

37. Secondary Outcome: Death Transcendence Scale
Description: 0-60 (higher score more death transcendence)
Time Frame: 2 weeks post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 33.98 (6.44) | 19.88 (6.41)

38. Secondary Outcome: Hopelessness
Description: 0-16 (higher score more hopeless)
Time Frame: 2 weeks post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 2.79 (0.76) | 6.08 (0.75)

39. Secondary Outcome: Hopelessness
Description: 0-16 (higher score more hopeless)
Time Frame: 26 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 2.30 (0.82) | 3.86 (0.82)

40. Secondary Outcome: Demoralization Scale
Description: 0-96 (higher score more demoralized)
Time Frame: 2-4 weeks prior to drug administration/ Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 35.71 (3.61) | 38.07 (3.49)

41. Secondary Outcome: Demoralization Scale
Description: 0-96 (higher score more demoralized)
Time Frame: 2 weeks post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 18.79 (3.61) | 32.79 (3.57)

42. Secondary Outcome: Demoralization Scale
Description: 0-96 (higher score more demoralized)
Time Frame: 26 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 19.38 (3.93) | 24.58 (3.92)

43. Secondary Outcome: QoL Physical Health Scale
Description: 4-20 (higher score improved quality of life domain)
Time Frame: 2-4 weeks prior to drug administration/ Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 15.14 (0.94) | 12.53 (0.91)

44. Secondary Outcome: QoL Physical Health Scale
Description: 4-20 (higher score improved quality of life domain)
Time Frame: 2 weeks post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 16.0 (0.94) | 12.44 (0.94)

45. Secondary Outcome: QoL Physical Health Scale
Description: 4-20 (higher score improved quality of life domain)
Time Frame: 26 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 16.77 (1.05) | 14.14 (1.05)

46. Secondary Outcome: QoL Psychological Scale
Description: 4-20 (higher score improved quality of life domain)
Time Frame: 2-4 weeks prior to drug administration/ Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 13.57 (.66) | 12.67 (.64)

47. Secondary Outcome: QoL Psychological Scale
Description: 4-20 (higher score improved quality of life domain)
Time Frame: 2 weeks post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 15.43 (.66) | 12.28 (.66)

48. Secondary Outcome: QoL Psychological Scale
Description: 4-20 (higher score improved quality of life domain)
Time Frame: 26 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 15.78 (.74) | 14.90 (0.74)

49. Secondary Outcome: QoL Social Relationships Scale
Description: 4-20 (higher score improved quality of life domain)
Time Frame: 2-4 weeks prior to drug administration/ Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 13.62 (.85) | 13.24 (.82)

50. Secondary Outcome: QoL Social Relationships Scale
Description: 4-20 (higher score improved quality of life domain)
Time Frame: 2 weeks post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 14.86 (.85) | 12.78 (.85)

51. Secondary Outcome: QoL Social Relationships Scale
Description: 4-20 (higher score improved quality of life domain)
Time Frame: 26 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 15.6 (.95) | 13.71 (.95)

52. Secondary Outcome: QoL Environment Scale
Description: 4-20 (higher score improved quality of life domain)
Time Frame: 2-4 weeks prior to drug administration/ Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 15.75 (.74) | 14.93 (.71)

53. Secondary Outcome: QoL Environment Scale
Description: 4-20 (higher score improved quality of life domain)
Time Frame: 2 weeks post drug administration 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 16.42 (0.74) | 13.90 (.74)

54. Secondary Outcome: QoL Environment Scale
Description: 4-20 (higher score improved quality of life domain)
Time Frame: 26 weeks post drug administration 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psilocybin First, Then Niacin | Niacin First, Then Psilocybin
Number analyzed (Participants) | 14 | 15
score on a scale | 16.96 (.82) | 15.82 (.82)

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Psilocybin; Niacin: Psilocybin and niacin will be administered in identically appearing opaque, size 0 gelatin capsules with approximately 180ml of water. The niacin dose will be 250mg
Arm/Group | Psilocybin | Niacin
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 1/29 | 0/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psilocybin (N=29) | Niacin (N=29)
Transient Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
elevations in BP and HR (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT00957359/Prot_SAP_000.pdf